CLINICAL TRIAL: NCT01946932
Title: Cognitive Impairment Following Cardiac Arrest and Target Temperature Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Copenhagen University Hospital, Denmark (Other); Azienda Ospedaliera Santa Maria Degli Angeli (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University Hospital of Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TTMcogsub
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-08

CONDITIONS: Heart Arrest; Out-of-hospital Cardiac Arrest; Cognition Disorders; Brain Injury
Keywords: Induced hypothermia; Mild induced hypothermia; Resuscitation; Therapeutic hypothermia; Neurological function; Cardiovascular diseases; Rehabilitation; Quality of life; Cognition
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Cognition Disorders; Brain Injuries; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac Arrest 33° (Active Comparator): survivors with temperature treatment 33°
  Interventions: Other: Temperature treatment
- Cardiac Arrest survivors 36° (Active Comparator): survivors with temperature treatment 36°
  Interventions: Other: Temperature treatment

INTERVENTIONS:
Other: Temperature treatment

SUMMARY:
This is a steering group approved substudy to the Target Temperature Management trial (TTM, ClinicalTrials.gov Identifier: NCT01020916). TTM compares the effect of two strictly controlled temperature regimes for survivors of out-of-hospital cardiac arrest.

The primary aim of this sub-study is to compare the amount of cognitive impairment in cardiac arrest survivors treated with 33 degrees and 36 degrees and with a matched group of control patients with myocardial infarction.

Our secondary aims are:

* To investigate the impact of cognitive impairment on our patients' ability to participate in society and their health related quality of life.
* To investigate the relationship between our patients cognitive impairments and their relatives/informants health related quality of life and feelings of burden.
* To test the hypothesis that the simple cognitive screening battery used in the TTM main trial is sensitive enough to detect all patients with significant cognitive disability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Out-of-Hospital Cardiac Arrest (OHCA)of presumed cardiac cause
* Unconsciousness after sustained return of spontaneous circulation (ROSC)

Exclusion Criteria at time for inclusion in the TTM study:

* Known bleeding diathesis
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed stroke
* Unwitnessed asystole
* Known limitations in therapy and Do Not Resuscitate-order
* Known disease making 180 days survival unlikely
* Known prearrest status Cerebral Performance Category (CPC)3 or 4
* Temperature <30°on admission

  * 4 hours (240 minutes) from ROSC to screening
* Systolic blood pressure <80 mm Hg in spite of fluid loading/vasopressor and/or inotropic medication/intra aortic balloon pump
* In-hospital cardiac arrest
* OHCA of presumed non-cardiac arrest cause

Additional Exclusion criteria for the sub-study:

* Disability to speak the site language well enough to complete tests without interpreter
* Controls should never have suffered a cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Rivermead Behavioural Memory Test (RBMT) | 180 days after Cardiac Arrest (CA) or Myocardial Infarction (MI)
  Memory test
Frontal Assessment Battery (FAB) | 180 days after CA or MI
  Screening of Executive functions
Symbol Digit Modalities Test (SDMT) | 180 days after CA or MI
  Assess attention, mental speed and concentration

SECONDARY OUTCOMES:
Mayo-Portland Adaptability Inventory-4 (MPAI-4) | 180 days after CA or MI
  Self rating of impairments, adjustment, and participation (in the society)
Short-Form Questionnaire 36 version 2 (SF-36v2) | 180 days after CA or MI
  Questionnaire of health-related quality of life, both for patient and informant/relative/caregiver
Zarit Burden Interview | 180 days after CA or MI
  Questionnaire for caregiver/informant/relative's perception of burden
Hospital Anxiety and Depression rating Scale (HADS) | 180 days after CA or MI
  Anxiety and Depression questionnaire
Two Simple Questions (TSQ) | 180 days after CA or MI
  Self rating of everyday activities and cognition
Informant Questionnaire on Cognitive Decline (IQCODE) | 180 days after CA or MI
  Patients cognitive functioning in everyday life, questionnaire completed by informant/relative/caregiver
MiniMental Status Examination (MMSE) | 180 days after CA or MI
  General cognitive screening
Cerebral Performance Category (CPC) | 180 days after CA or MI
  Scale for general neurological outcome
modified Rankin Scale | 180 days after CA or MI
  Scale for general outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Cronberg, MD, PhD, Study Chair — Department of Clinical Sciences, Lund University, Lund, Sweden and Department of Neurology, Skåne University Hospital, Lund, Sweden; Niklas Nielsen, MD,PhD, Principal Investigator — Department of Clinical Sciences, Lund University, Lund Sweden and Department of Anesthesia and Intensive Care, Helsingborg Hospital, Helsingborg, Sweden; Jesper Kjaergaard, MD, PhD, Principal Investigator — The Heart Centrem Copenhagen University, Copenhagen, Denmark; Janneke Horn, MD, PhD, Principal Investigator — Department of Intensive Care, Academic Medical Centrum, Amsterdam, Netherlands; Tommaso Pellis, MD, PhD, Principal Investigator — Intensive Care Unit Santa Maria Degli Angeli, Pordenonde, Italy; Matthew P Wise, MD, PhD, Principal Investigator — Adult Critical Care, University Hospital of Wales, Cardiff, Untied Kingdom; Gisela Lilja, OT, Study Director — Lund University Hospital, Lund, Sweden
Locations (20):
- Rigshospitalet, Copenhagen, Denmark
- Italy (3):
  - San Martino Hospital, Genova
  - Santa Maria degli Angeli Hospital, Pordenone
  - Ospedale Universitario di Cattinaria, Trieste
- Netherlands (4):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Leeuwarden Hospital, Leeuwarden
- Sweden (8):
  - Sahlgrenska University Hospital, Thorax, Gothenburg
  - Sahlgrenska University Hospital, Östra, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Karlstad Central Hospital, Karlstad
  - Skåne University Hospital, Lund, Lund
  - Skåne University Hospital, Malmö, Malmo
  - Örebro University Hospital, Örebro
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - St Georges' Hospital, London
  - Royal Berkshire NHS Foundation Trust, Reading

REFERENCES:
- [Background] Cronberg T, Lilja G, Rundgren M, Friberg H, Widner H. Long-term neurological outcome after cardiac arrest and therapeutic hypothermia. Resuscitation. 2009 Oct;80(10):1119-23. doi: 10.1016/j.resuscitation.2009.06.021. Epub 2009 Jul 23. PMID 19631442
- [Background] Nielsen N, Wetterslev J, al-Subaie N, Andersson B, Bro-Jeppesen J, Bishop G, Brunetti I, Cranshaw J, Cronberg T, Edqvist K, Erlinge D, Gasche Y, Glover G, Hassager C, Horn J, Hovdenes J, Johnsson J, Kjaergaard J, Kuiper M, Langorgen J, Macken L, Martinell L, Martner P, Pellis T, Pelosi P, Petersen P, Persson S, Rundgren M, Saxena M, Svensson R, Stammet P, Thoren A, Unden J, Walden A, Wallskog J, Wanscher M, Wise MP, Wyon N, Aneman A, Friberg H. Target Temperature Management after out-of-hospital cardiac arrest--a randomized, parallel-group, assessor-blinded clinical trial--rationale and design. Am Heart J. 2012 Apr;163(4):541-8. doi: 10.1016/j.ahj.2012.01.013. PMID 22520518
- [Derived] Heimburg K, Cronberg T, Tornberg AB, Ullen S, Friberg H, Nielsen N, Hassager C, Horn J, Kjaergaard J, Kuiper M, Rylander C, Wise MP, Lilja G. Self-reported limitations in physical function are common 6 months after out-of-hospital cardiac arrest. Resusc Plus. 2022 Jul 19;11:100275. doi: 10.1016/j.resplu.2022.100275. eCollection 2022 Sep. PMID 36164471
- [Derived] Lilja G, Nielsen N, Bro-Jeppesen J, Dunford H, Friberg H, Hofgren C, Horn J, Insorsi A, Kjaergaard J, Nilsson F, Pelosi P, Winters T, Wise MP, Cronberg T. Return to Work and Participation in Society After Out-of-Hospital Cardiac Arrest. Circ Cardiovasc Qual Outcomes. 2018 Jan;11(1):e003566. doi: 10.1161/CIRCOUTCOMES.117.003566. PMID 29326145
- [Derived] Lilja G, Nilsson G, Nielsen N, Friberg H, Hassager C, Koopmans M, Kuiper M, Martini A, Mellinghoff J, Pelosi P, Wanscher M, Wise MP, Ostman I, Cronberg T. Anxiety and depression among out-of-hospital cardiac arrest survivors. Resuscitation. 2015 Dec;97:68-75. doi: 10.1016/j.resuscitation.2015.09.389. Epub 2015 Oct 9. PMID 26433116
- [Derived] Lilja G, Nielsen N, Friberg H, Horn J, Kjaergaard J, Nilsson F, Pellis T, Wetterslev J, Wise MP, Bosch F, Bro-Jeppesen J, Brunetti I, Buratti AF, Hassager C, Hofgren C, Insorsi A, Kuiper M, Martini A, Palmer N, Rundgren M, Rylander C, van der Veen A, Wanscher M, Watkins H, Cronberg T. Cognitive function in survivors of out-of-hospital cardiac arrest after target temperature management at 33 degrees C versus 36 degrees C. Circulation. 2015 Apr 14;131(15):1340-9. doi: 10.1161/CIRCULATIONAHA.114.014414. Epub 2015 Feb 13. PMID 25681466
- [Derived] Lilja G, Nielsen N, Friberg H, Horn J, Kjaergaard J, Pellis T, Rundgren M, Wetterslev J, Wise MP, Nilsson F, Cronberg T. Cognitive function after cardiac arrest and temperature management; rationale and description of a sub-study in the Target Temperature Management trial. BMC Cardiovasc Disord. 2013 Oct 12;13:85. doi: 10.1186/1471-2261-13-85. PMID 24118853